CLINICAL TRIAL: NCT03573518
Title: A Randomized, Double-Blind, Vehicle-Controlled Study to Evaluate the Safety and Efficacy of BTX 1503 in Patients With Moderate to Severe Acne Vulgaris
Brief Title: Evaluation of BTX 1503 in Patients With Moderate to Severe Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Botanix Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTX.2018.001
Record Dates: First submitted 2018-06-19; First posted 2018-06-29 (Actual); Results first posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Acne Vulgaris
Keywords: Synthetic CBD; Cannabidiol
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- BTX 1503 5% BID (Experimental): BTX 1503 5% CBD (w/w) solution twice daily
  Interventions: Drug: BTX 1503
- BTX 1503 5% QD (Experimental): BTX 1503 5% CBD (w/w) solution once daily
  Interventions: Drug: BTX 1503
- BTX 1503 2.5% QD (Experimental): BTX 1503 2.5% CBD (w/w) solution once daily
  Interventions: Drug: BTX 1503
- Vehicle BID (Placebo Comparator): Vehicle twice daily
  Interventions: Drug: Vehicle
- Vehicle QD (Placebo Comparator): Vehicle once daily
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: BTX 1503 — BTX 1503 Dose 1 liquid formulation, or BTX 1503 Dose 2 liquid formulation
  Other Names: BTX1503
  Arms: BTX 1503 2.5% QD; BTX 1503 5% BID; BTX 1503 5% QD
Drug: Vehicle — Placebo
  Arms: Vehicle BID; Vehicle QD

SUMMARY:
The objective of this study is to assess safety and efficacy of various doses of BTX 1503 liquid formulation in subjects with moderate to severe acne vulgaris of the face.

DETAILED DESCRIPTION:
This will be a multi-center, randomized, double-blinded, vehicle-controlled, parallel group, dose-finding study in pediatrics, adolescents and adults (aged 12 to 40 years). The objective of this study is to assess the safety and efficacy of various doses of BTX 1503 in subjects with moderate to severe acne vulgaris of the face.

ELIGIBILITY:
Inclusion Criteria:

1. Subject (or legal guardian) has the ability and willingness to sign a written informed consent/assent.
2. Subject is of either gender and 12 to 40 years of age.
3. Subject is in good general health without clinically significant haematological, cardiac, respiratory, renal, endocrine, gastrointestinal, psychiatric, hepatic, or malignant disease, as determined by the investigator.
4. Subject has suitable venous access for blood sampling.
5. Subject is able and willing to complete the study and to comply with all study instructions and attend the necessary visits.
6. Subject has acne vulgaris of the face defined as:

   1. 20 to 50 (inclusive) inflammatory lesions on the face
   2. 20 to 100 (inclusive) non-inflammatory lesions on the face
   3. An Investigator's Global Assessment (IGA) score for acne severity of 3 or 4 (moderate or severe) assessed on the face.
7. Subject has ≤ 2 nodular/cystic acne lesions (>5 mm in diameter).
8. Subject must refrain from the use of other treatments for acne during the study.
9. Subject must agree to not wash or shave their face, swim or otherwise get their face wet for at least 1 hour after application of study medication.
10. Subject must agree to maintain their regular use of sunscreens, moisturizers, shaving cream, and facial make up throughout the entire course of the study.
11. Male subjects and their partners must agree and commit to use a barrier method of contraception during the study and for 90 days after last study drug application.
12. A negative UPT result for all WOCBP at the Screening Visit and Baseline Visit, if applicable. A WOCBP is one who is not permanently sterilized or is not postmenopausal. Postmenopausal is defined as 24 months with no menses without an alternative medical cause.
13. Sexually active women must agree to use the following throughout the study and for 30 days after last study drug application:

    a. One of these highly effective contraception methods i. Intrauterine device (IUD); hormonal (injections, implants, transdermal patch, vaginal ring; tubal ligation; partner vasectomy, OR b. Oral contraceptives WITH a barrier method (listed below), OR c. Two barrier forms of contraception (listed below) i. Male or female condom; diaphragm; cervical cap.
14. Male subjects must refrain from sperm donation during the study treatment period until 90 days after final study drug administration.
15. Male subjects must agree to keep their face clean shaven (no moustache or goatee; short sideburns acceptable) throughout the study and use the same method for shaving as was used for the 4 weeks prior to the Screening Visit.

Exclusion Criteria:

1. People who would otherwise qualify for the study but are living in the same household as a study subject, are not allowed to participate in the study.
2. Female subject who is breast feeding, pregnant, or planning to become pregnant any time during the course of the study.
3. Subject with history of known or suspected intolerance to the drug product excipients.
4. Subject has known HIV infection.
5. Subject has acne conglobata, acne fulminans, secondary acne (chloracne), pseudo-folliculitis, severe acne requiring systemic treatment, or is taking a medication known to induce or exacerbate acne.
6. Subject has severe truncal acne.
7. Subject has excessive facial hair that would interfere with the evaluation of safety or with the diagnosis or assessment of acne vulgaris.
8. Subject has sunburns, unevenness in skin tones, tattoos, scars, excessive hair, freckles, birthmarks, moles, or other skin damage or abnormality that would result in the inability to evaluate the skin of the face.
9. Subject has any skin condition of the face other than acne vulgaris.
10. Subject has used oral retinoid (e.g. isotretinoin) within 6 months (180 days) prior to the Baseline Visit.
11. Subject has used Vitamin A supplements greater than 10,000 units/day within 6 months (180 days) prior to the Baseline Visit.
12. Subject has used androgen receptor blockers (such as spironolactone or flutamide) within 3 months (90 days) prior to the Baseline Visit.
13. Subject has initiated treatment with hormonal therapy or changed dosing with hormonal therapy within 3 months (90 days) prior to the Baseline Visit.
14. Subject has had facial procedures (chemical or laser peel, microdermabrasion, etc.) within 8 weeks (56 days) prior to the Baseline Visit.
15. Subject has had treatment with systemic antibiotics within 4 weeks (28 days) prior to the Baseline Visit.
16. Subject has had treatment with systemic anti-acne drugs within 4 weeks (28 days) prior to the Baseline Visit.
17. Subject has had treatment with systemic anti-inflammatory drugs within 4 weeks (28 days) prior to the Baseline Visit.
18. Subject has had treatment with systemic (oral) corticosteroids other immunosuppressive medications within 4 weeks (28 days) prior to the Baseline Visit.
19. Subject has had treatment with prescription topical retinoid use on the face (e.g. tretinoin, tazarotene) within 4 weeks (28 days) prior to the Baseline Visit.
20. Subject has had treatment with topical prescription antibiotics (e.g. dapsone, clindamycin, erythromycin, or sulfacetamide) or combination products that include a topical antibiotic within 2 weeks (14 days) prior to the Baseline Visit.
21. Subject has had treatment with over-the-counter (OTC) topical medications for the treatment of acne vulgaris including benzoyl peroxide, topical anti- inflammatory medications, corticosteroids, adapalene, α-hydroxy/glycolic acid on the face within 2 weeks (14 days) prior to the Baseline Visit.
22. Subject is currently using any medication that, in the opinion of the investigator, may affect the evaluation of the study product or place the subject at undue risk.
23. Subject has had photodynamic therapy within 8 weeks (56 days) prior to the Baseline Visit.
24. Subject has used a tanning bed within 2 weeks (14 days) prior to the Baseline Visit.
25. Subject has used home-based light treatment within 2 weeks (14 days) prior to the Baseline Visit.
26. Subject has an underlying disease that requires the use of interfering topical or systemic therapy.
27. Subject has other dermatological conditions that require the use of interfering topical or systemic therapy or that might interfere with study assessments such as, but not limited to, atopic dermatitis, psoriasis, perioral dermatitis, or rosacea.
28. Subject has had excessive sun exposure (in the opinion of the investigator) within one week prior to the Baseline Visit and an unwillingness to refrain from excessive sun exposure during the study.
29. Subject has a clinically relevant history or currently suffering from any disease or condition that, in the opinion of the investigator, may affect the evaluation of the study product or place the subject at undue risk. This may include respiratory (including chronic asthma requiring repetitive drug interventions), gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, or connective tissue diseases or disorders.
30. Subject has a clinically relevant history of, or current evidence of, abuse of alcohol or other drugs. Subjects may be deemed eligible if the UDS identifies subject-reported, prescribed drugs or appropriate levels of alcohol, as determined by the investigator.
31. Subject has participated in another investigational drug or device research study within 4 weeks (28 days) of the Baseline Visit or five half-lives of the drug, whichever is longer.
32. Any other reason that would make the subject, in the opinion of the investigator or sponsor, unsuitable for the study.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 368 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Robinson, CRNP, Study Director — Head of Development, Botanix Pharmaceuticals
Locations (36):
- United States (25):
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Encino Research Center, Encino, California
  - Dermatology Specialist, Inc., Murrieta, California
  - Quest Dermatology Research, Northridge, California
  - Clinical Science Insitute, Santa Monica, California
  - Well Phrama Medical Research, Miami, Florida
  - Tory Sullivan, M.D., PA, North Miami Beach, Florida
  - Precision Clinical Research, Sunrise, Florida
  - DS Research - Louisville, Louisville, Kentucky
  - Delricht Research, New Orleans, Louisiana
  - Metro Boston Clinical, Brighton, Maine
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Medisearch Clinical Trials, Saint Joseph, Missouri
  - Washington University School of Medicine - Dermatology, St Louis, Missouri
  - JDR Dermatology Research, Las Vegas, Nevada
  - The Acne Treatment and Research Center, Morristown, New Jersey
  - Aventiv Research, Dublin, Ohio
  - Penn State Hershey Medical, Hershey, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Greenville Dermatology, LLC, Greenville, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Avant Research Associates, LLC, Austin, Texas
  - DermReasearch, Austin, Texas
  - J&S Studies, Inc., College Station, Texas
  - Suzanne Bruce and Associates, PA, Houston, Texas
- Australia (11):
  - Cmax Clinical Research, Adelaide
  - The Skin Centre, Benowa
  - Burswood Dermatology, Burwood
  - Skin & Canver Foundation Inc., Carlton
  - Sinclair Dermatology, East Melbourne
  - Fremantle Dermatology, Fremantle
  - North Eastern Health Specialist, Hectorville
  - St George Dermatology & Skim Cancer Center, Kogarah
  - Captain Sterline Medical Centre, Nedlands
  - Woden Dermatology, Phillip
  - Varacity Clinical Research, Woolloongabba

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vehicle Combined (BID or QID): Placebo BID + Placebo QD
  =Placebo Combined group
Period: Overall Study
Arm/Group | BTX 1503 5% BID | BTX 1503 5% QD | BTX 1503 2.5% QD | Vehicle Combined (BID or QID)
Started | 92 | 92 | 92 | 92
Completed | 69 | 77 | 70 | 81
Not Completed | 23 | 15 | 22 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BTX 1503 5% BID | BTX 1503 5% QD | BTX 1503 2.5% QD | Vehicle Combined (BID or QID) | Total
Number analyzed (Participants) | 92 | 92 | 92 | 92 | 368
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.5 (6.65) | 19.7 (5.99) | 19.4 (5.98) | 20.5 (6.14) | 20.0 (6.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 60 | 58 | 55 | 229
  Male | 36 | 32 | 34 | 37 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 21 | 23 | 23 | 93
  Not Hispanic or Latino | 66 | 71 | 69 | 69 | 275
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 5 | 5 | 5 | 7 | 22
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 1 | 1 | 5
  Black or African American | 12 | 5 | 5 | 6 | 28
  White | 67 | 75 | 73 | 72 | 287
  More than one race | 5 | 6 | 8 | 6 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Inflammatory Lesion Count [Mean (Standard Deviation); unit: Lesions] | 29.3 (8.52) | 28.5 (8.95) | 29.6 (8.00) | 29.1 (8.25) | 29.1 (8.37)

OUTCOME MEASURES:

1. Primary Outcome: Safety as Measured by Reported Adverse Events
Description: Summary of Treatment-Emergent Adverse Events by MedDra Preferred Term that Occurred with a Frequency > 2% in any Treatment Group (Safety Population)
Time Frame: Day 84
Population: Safety Population
Measure: Number; unit: TEAEs
Arm/Group | BTX 1503 5% BID | BTX 1503 5% QD | BTX 1503 2.5% QD | Vehicle Combined (BID or QID)
Number analyzed (Participants) | 92 | 91 | 91 | 91
TEAEs
  Upper Respiratory tract infection | 2 | 4 | 5 | 5
  Viral upper respiratory tract infection | 3 | 2 | 3 | 4
  Headache | 1 | 1 | 2 | 0
  Acne | 2 | 0 | 2 | 0
  Cough | 1 | 0 | 2 | 0
  Oropharyngeal pain | 0 | 2 | 0 | 1

2. Secondary Outcome: Absolute Change From Baseline in Inflammatory Lesion Counts
Description: Summary of Absolute Change from Baseline in Inflammatory Count at Day 84 (Intent-to-Treat Population)
Time Frame: Day 84
Population: Intent-to-Treat Population
Measure: Least Squares Mean (Standard Deviation); unit: Lesions
Arm/Group | BTX 1503 5% BID | BTX 1503 5% QD | BTX 1503 2.5% QD | Vehicle Combined (BID or QID)
Number analyzed (Participants) | 92 | 92 | 91 | 92
Lesions | -8.5 (12.57) | -12 (12.58) | -11.7 (12.57) | -11.3 (12.57)

ADVERSE EVENTS:
Time Frame: Approximately 3 months
Description: Reporting of AE's included reporting of pregnancy
Arm/Group | BTX 1503 5% BID | BTX 1503 5% QD | BTX 1503 2.5% QD | Vehicle Combined (BID or QID)
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/91 | 0/91 | 0/91
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/91 | 0/91 | 0/91
Other Adverse Events (participants affected / at risk) | 9/92 | 9/91 | 14/91 | 10/91
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BTX 1503 5% BID (N=92) | BTX 1503 5% QD (N=91) | BTX 1503 2.5% QD (N=91) | Vehicle Combined (BID or QID) (N=91)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 5 (5) | 5 (5)
Viral upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Oorpharyngeal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
As Study is a Multi-centre Study, no Publication of the Study results may be made until Publication of the results of the Multi-centre study or 2 years after Study Completion, whichever is sooner.

DOCUMENTS (2):
  • Study Protocol (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/18/NCT03573518/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT03573518/SAP_001.pdf